CLINICAL TRIAL: NCT03873519
Title: Acute Effect of Chromatic Environment During Chemotherapy Sessions on Health Status and Pain
Brief Title: Acute Effect of Chromatic Environment During Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Instituto Oncológico Balselga (Unknown)
Responsible Party: Principal Investigator, Margarita Perez, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-2017/UEM11
Record Dates: First submitted 2018-09-11; First posted 2019-03-13 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: chemotherapy; vital signs; stress; health status; healing environment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be allocated into four conditions (Group A: Cold North, Group B: Cold South C: Warm North D: Warm South), and they will be assigned a new condition at each next visit. The sequence will be assigned randomly to each patient. During each of the four visits, the patients will be treated per standard of care during their chemotherapy sessions. Outcome variables will be assessed before and after each visit.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold North (Experimental): Group A: Cold color scheme, room facing North
  Interventions: Other: Chromatic Environment; Other: Room Orientation
- Cold South (Experimental): Group B:Cold color scheme, room facing South
  Interventions: Other: Chromatic Environment; Other: Room Orientation
- Warm North (Experimental): Group C: Warm color scheme, room facing North
  Interventions: Other: Chromatic Environment; Other: Room Orientation
- Warm South (Experimental): Group D: Warm color scheme, room facing South
  Interventions: Other: Chromatic Environment; Other: Room Orientation

INTERVENTIONS:
Other: Chromatic Environment — Rooms where chemotherapy sessions are delivered will be modified to show warm/cold color temperature in walls and equipment.
Other: Room Orientation — Room will be facing North or South

SUMMARY:
The primary objective is to examine the acute effect of color, room orientation (affecting amount of luminosity) on perceived health status and stress levels in oncologic patients during chemotherapy sessions at outpatient clinic. The secondary objectives will be to study the effect on vital signs (body temperature, heart rate, systolic blood pressure). Patients will be allocated into four conditions (Group A: Cold North, Group B: Cold South C: Warm North D: Warm South) for each session. For the next session, patients will be assigned a new condition. Assignment of sequences will be randomized for each patient.

20 patients will be randomly assigned to one of the four groups, after having signed the Free and Informed Consent Form and agreed to participate in the project, will respond to the evaluation form and will be submitted to physical examination. Patients will be treated per standard of care.

ELIGIBILITY:
Inclusion criteria:

* Age 18-89 years
* Diagnosed with breast cancer that required chemotherapy
* Followed in outpatient clinic

Exclusion criteria:

* Diagnosed color blindness
* Undergoing treatment with antidepressants

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
EUROQOL-5D-5L questionnaire: Mobility | 5 minutes before to 5 minutes after chemotherapy session
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement using a 1-digit number that expresses the level selected for that dimension.
EUROQOL-5D-5L questionnaire: Self-care | 5 minutes before to 5 minutes after chemotherapy session
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement using a 1-digit number that expresses the level selected for that dimension.
EUROQOL-5D-5L questionnaire: Usual activities | 5 minutes before to 5 minutes after chemotherapy session
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement using a 1-digit number that expresses the level selected for that dimension.
EUROQOL-5D-5L questionnaire: Pain/Discomfort | 5 minutes before to 5 minutes after chemotherapy session
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement using a 1-digit number that expresses the level selected for that dimension.
EUROQOL-5D-5L questionnaire: Anxiety/Depression | 5 minutes before to 5 minutes after chemotherapy session
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement using a 1-digit number that expresses the level selected for that dimension.
EUROQOL-5D-5L questionnaire: EQ-VAS | 5 minutes before to 5 minutes after chemotherapy session
  The EQ VAS is an independent subscale of the EUROQOL-5D-5L questionnaire, which uses a vertical visual analogue scale format. The EQ VAS is used for recording the self-rated health on a range from 0 to 100, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement

SECONDARY OUTCOMES:
ID-Pain questionnaire | 5 minutes before to 5 minutes after chemotherapy session
  Assessment of neuropathic pain
Vital signs: body temperature | 5 minutes before to 5 minutes after chemotherapy session
  Per standard of care, in Celsius
Vital signs: blood pressure | 5 minutes before to 5 minutes after chemotherapy session
  Per standard of care, in mm Hg
Vital signs: heart rate | 5 minutes before to 5 minutes after chemotherapy session
  Per standard of care, in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Pérez Ruiz, MD, PhD, Study Chair — Universidad Europea
Locations (1):
- Hospital Ruber Internacional, Madrid, Spain

REFERENCES:
- [Derived] Gomez-Vela P, Perez-Ruiz M, Hernandez Martin MF, Roman J, Larumbe-Zabala E. Acute effect of orange chromatic environment on perceived health status, pain, and vital signs during chemotherapy treatment. Support Care Cancer. 2020 May;28(5):2321-2329. doi: 10.1007/s00520-019-05064-w. Epub 2019 Sep 3. PMID 31482404